CLINICAL TRIAL: NCT07192393
Title: Quantifying the Household Impact on Patient-Reported Outcomes and Costs Associated With the Care of Preterm Babies With and Without Necrotising Enterocolitis (NEC): A Study Alongside the Withholding Enteral Feeds Around Blood Transfusion (WHEAT) Trial
Brief Title: Health-Related Quality-of-Life and Household Financial and Wellbeing Impacts of Prematurity and Necrotising Enterocolitis (NEC).
Acronym: PREM-IMPACT
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Oxford (Other); University of Leeds (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Other Study IDs: 351166
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Prematurity; Extreme; Prematurity; Decision Support; Necrotising Enterocolitis; Preterm; Preterm Birth; Preterm Infant Health
Keywords: NEC; Cost-Effectiveness Analysis; Cost-Utility Analysis; Health-Related Quality of Life; HR-QoL; Prematurity; Preterm; Health Economic Analysis; Financial Impact; Wellbeing
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Prematurity: Includes all babies born <30 weeks gestation, who did not develop NEC during their hospital stay, and their parents and siblings.
- General Prematurity + Necrotising Enterocolitis (NEC): Includes all babies born <30 weeks gestation, who also developed and recovered from NEC during their hospital stay, and their parents and siblings.

SUMMARY:
PREM-IMPACT is a UK-based observational study exploring how caring for a very premature baby-particularly one affected by necrotising enterocolitis (NEC)-impacts families over the first year after hospital discharge. NEC is a serious bowel disease that can occur in premature babies, often requiring surgery and prolonged hospitalisation.

This study runs alongside the WHEAT International Trial, which investigates whether pausing or continuing milk feeds during blood transfusions affects the risk of NEC in very preterm babies. PREM-IMPACT acts as a nested economic evaluation of the WHEAT Trial, helping to understand whether different feeding practices around transfusion offer good value for money from both the NHS and family perspective.

PREM-IMPACT will collect detailed data on babies' health-related quality of life, as well as the financial, emotional, and social impact on parents and siblings. Families are recruited from neonatal units when their baby is ready to go home and complete questionnaires at three timepoints: 1) just before discharge, 2) six months later, and 3) twelve months later. Questionnaires cover health, wellbeing, healthcare use, and costs to the family (such as travel, time off work, or extra care needs). A dedicated research nurse based at the lead NHS site helps coordinate follow-up centrally.

By studying families of babies with and without NEC, this project aims to clarify the burden of prematurity and NEC on infant outcomes and family wellbeing. The results will inform future policy decisions, including whether pausing or continuing milk feeds during transfusion should be adopted in routine neonatal care.

DETAILED DESCRIPTION:
PREM-IMPACT (PREMaturity IMPACT): Quantifying the Household Impact on Patient-Reported Outcomes and Costs Associated with the Care of Preterm Babies with and without Necrotising Enterocolitis (NEC): A Study alongside the WHEAT Trial

Background Necrotising enterocolitis (NEC) is a severe gastrointestinal condition affecting very preterm infants, associated with high mortality and significant long-term morbidity. Despite progress in neonatal care, NEC remains a major contributor to healthcare burden and family distress. The WHEAT International Trial is evaluating whether pausing vs continuing enteral feeds during packed red cell transfusion influences NEC incidence in very preterm infants. However, an economic evaluation was not built into WHEAT due to funding limitations.

Study Design PREM-IMPACT is a prospective, observational cohort study embedded within UK sites participating in the WHEAT Trial. Its aim is to quantify the household and health system impacts associated with NEC and evaluate the cost-effectiveness of feeding practices during transfusion. This includes examining infant health-related quality of life (HRQoL), parental and sibling wellbeing, healthcare resource use, and economic burden to families and the NHS.

Recruitment A minimum of 75 families of babies born at <30 weeks' gestation will be recruited from neonatal units across 5-7 NHS hospitals. Families will be stratified by NEC diagnosis (NEC vs no NEC). Data collection occurs at three timepoints: baseline (just prior to neonatal discharge), 6 months post-discharge, and 12 months post-discharge.

Data

Data collected in the study include:

* Infant clinical information (birth, diagnoses, feeding method, length of stay)
* Parental and sibling demographics
* Infant HRQoL (EQ-TIPS, parent proxy)
* Parent HRQoL and wellbeing (EQ-5D-5L, EQ-HWB, ICECAP-A)
* Sibling HRQoL (EQ-TIPS or EQ-5D-Y, depending on age)
* Financial impact (out-of-pocket expenses, income loss, employment changes)
* Healthcare utilisation (readmissions, outpatient visits, GP visits, therapies)

Analyses Descriptive and comparative analyses will explore group differences in costs and outcomes. Quality-adjusted life years (QALYs) will be derived for each family member using appropriate value sets. A cost-consequence analysis will be performed to assess the overall burden of NEC. In addition, cost and utility data collected in PREM-IMPACT will be combined with clinical effectiveness data from infants enrolled in the WHEAT International Trial to conduct a model-based cost-effectiveness analysis (CEA) of feeding practices during transfusion. The CEA will adopt both NHS and societal perspectives.

Impact This study addresses a critical evidence gap by capturing the broader health and financial consequences of NEC and prematurity across the family unit. Findings will inform future resource allocation and neonatal care policy decisions.

ELIGIBILITY:
Inclusion Criteria:

* Preterm birth <30 gestational weeks

Exclusion Criteria:

* Parent(s) of a preterm baby who died of necrotising enterocolitis (NEC)
* Parent(s) unwilling or unable to provide written informed consent
* Parent(s) and sibling(s) unable to understand English.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of 90 babies will be recruited.
  We have identified at least 9 high-volume recruiting sites for the WHEAT International trial, including 3 regional neonatal surgical units. These sites collectively care for over 300 eligible babies and over 100 babies with NEC annually. Our site selection ensures a diverse sample of parents, representing various socioeconomic and ethnic backgrounds, with all sites located in areas of both affluence and deprivation.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Infant Health-Related Quality of Life (HRQoL) | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Parent-reported proxy measure of infant HRQoL using the EQ-TIPS questionnaire, completed at discharge, 6 months, and 12 months post-discharge.
Infant Healthcare Resource Utilisation | At 6 months post-neonatal discharge and 12 months post-neonatal discharge.
  Number and type of healthcare services used by the infant over the first year following neonatal discharge, including hospital readmissions, outpatient visits, emergency visits, primary care, and additional medical interventions related to NEC or prematurity.
Household Financial Impact | At 6 months post-neonatal discharge and 12 months post-neonatal discharge.
  Out-of-pocket costs, time off work, and financial strain experienced by parents or caregivers, captured using a study-specific questionnaire at 6 and 12 months.

SECONDARY OUTCOMES:
Parental Health-Related Quality of Life | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Self-reported HRQoL of parents using EQ-5D-5L at three timepoints.
Parental Wellbeing Capabilities | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Self-reported wellbeing scores using EQ-HWB instruments
Sibling Health-Related Quality of Life (EQ-TIPS, ages 0-3) | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Proxy-reported HRQoL of siblings aged 0-3 years using the EQ-TIPS instrument.
Economic Evaluation of the WHEAT International Trial | From study start through study completion, approximately 2 years.
  Cost-effectiveness analysis (CEA) of continue vs pause feeds during routine packed red cell transfusion. Summary of cost and utilities collected from this study, to clinical effectiveness from matched participants (babies) enrolled in the WHEAT international trial.
Parental Wellbeing Capabilities | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Self-reported wellbeing (capability) scores using ICECAP-A instruments.
Sibling Health-Related Quality of Life (EQ-5D-Y-3L, ages 4-15) | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Age-appropriate self- or proxy-reported HRQoL of siblings aged 4-15 years using the EQ-5D-Y-3L instrument.
Sibling Health-Related Quality of Life (EQ-5D-5L, ages 16+) | Baseline (at the point of discharge home from neonatal care), 6 months post-neonatal discharge, and 12 months post-neonatal discharge.
  Age-appropriate self- or proxy-reported HRQoL of siblings aged 16+ years using the EQ-5D-5L instrument.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University Hospital Coventry, Coventry
  - Liverpool Women's Hospital, Liverpool
  - Chelsea & Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No